CLINICAL TRIAL: NCT07095881
Title: Peri-implant Soft Tissue Response to Direct Zirconia-Based Composite Customized Healing Abutment: A Randomized Controlled Clinical Study With Biochemical Analysis
Brief Title: Peri-implant Soft Tissue Response to Direct Zirconia-Based Composite Customized Healing Abutment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, ahmed asem elsayed abd elmoteleb, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-REC 1437
Record Dates: First submitted 2025-07-16; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Missing Tooth
Keywords: Implant; dental implant; Delayed implant; Healing abutment; Customized healing abutment; Zirconia-based composite customized healing abutment; Conventional composite customized healing abutment; Biochemical Analysis; Pink esthetic Score; Papilla index; PISF samples; IL-1β
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel design, two arms clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia-based composite customized healing abutment (Active Comparator): Participants in this arm will receive a customized healing abutment made of Zirconia-based composite material fabricated chairside.
  The abutment will be designed to mimic the emergence profile of the final prosthesis, aiming to optimize soft tissue shaping and healing.
  The abutment is placed immediately after implant placement and will remain in place for 3 months.
  Interventions: Other: Zirconia-based composite customized healing abutment
- Conventional composite customized healing abutment (Active Comparator): Participants in this arm will receive a customized healing abutment made of conventional composite material fabricated chairside.
  The abutment will be designed to mimic the emergence profile of the final prosthesis, aiming to optimize soft tissue shaping and healing.
  The abutment is placed immediately after implant placement and will remain in place for 3 months.
  Interventions: Other: Conventional composite customized healing abutment.

INTERVENTIONS:
Other: Zirconia-based composite customized healing abutment — using Zirconia-based composite in customized healing abutment fabrication
  Arms: Zirconia-based composite customized healing abutment
Other: Conventional composite customized healing abutment. — using conventional composite in customized healing abutment fabrication
  Arms: Conventional composite customized healing abutment

SUMMARY:
The goal of this clinical trial is to learn if using zirconia-based composite customized healing abutment can have a favorable effect on peri implant soft tissue that may be related to the superior biological properties of zirconium nano particles regarding increased biocompatibility and decreased inflammatory response Patients that are eligible for implant placement

The main question it aims to answer is:

Does zirconia-based composite customized healing abutment have a significantly different effect on peri-implant soft tissue compared to conventional composite customized healing abutment in terms of biological properties or biocompatibility or inflammatory response? Researchers will compare between direct zirconia-based composite customized healing abutments vs conventional composite customized healing abutments placed simultaneously with delayed dental implant placement.

Participants will be undergo the following procedures :

A) Presurgical procedures:

1. Detailed clinical examination, full history, and radiographic examination (CBCT) will be performed initially to aid in patients' selection.
2. After enrollment, all participants will sign the informed consent.
3. All participants will be subjected to periodontal phase I treatment including periodontal supra- and sub-gingival debridement and oral hygiene instructions.

B) Surgical procedures:

1. After local anesthesia administration, flap is raised, osteotomy site preparation, and implant will be placed.
2. Check the ISQ to exceed or equal 70 unit.
3. A customized Light-cured Direct Zirconia-Based Composite or A customized Light-cured Direct Convential Composite Healing Abutment will be placed.

Then all participants should follow up at the following times : Baseline, 1,2 and 3 months after implantation.

DETAILED DESCRIPTION:
Light-cured direct zirconia-based composite has many potential uses in dentistry, because of mechanical and biological reasons maintaining the health of peri-implant soft tissues during healing.

Direct zirconia-based composite customized healing abutments have superior properties such as biocompatibility, chemical stability, antibacterial and mechanical properties.

Aim of the study: This study will be carried out to compare zirconia-based composite customized healing abutments vs conventional composite customized healing abutment placed simultaneously with delayed dental implant placement.

Materials and Methods: This will be done by clinical evaluation of peri-implant soft tissue changes. Moreover, peri-implant sulcus fluid (PISF) will be measured for the level of Interleukin-1 beta (IL-1β) in the gingival crevicular fluid.

PICOTS Elements:

Patient/Problem:Patients that are eligible for implant placement within inclusion criteria.

Intervention: Zirconia-based composite customized healing abutment. Comparator: Conventional composite customized healing abutment.

Outcome:

Primary outcome : Clinical evaluation of peri-implant soft tissue changes via pink esthetic score and papilla index.

Secondary outcome : Biochemical assessment of IL-1β level in the gingival crevicular fluid using Periopaper strip .

Time: Baseline, 1,2 and 3 months after implantation. Biochemical assessment : after 2 months of implantation. Setting: Faculty of Dentistry, Ain Shams University. Clinical Relevance: The result will affect the gold standard in choosing the customized healing abutment material for implant patients, regarding which one offers better peri-implant soft tissue results, healing stimulation, and less inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be systematically free from any disease as according to Cornell Medical Index-Health Questionnaire (Pendleton et al., 2004).
2. Both genders.
3. Age from 20-50 years.
4. Missing tooth to be restored with standard implant, with no need for additional bone and soft tissue augmentation procedures (Beretta et al., 2019).
5. Implants primary stability ISQ ≥ 70 unites using the Osstell Mentor (Baltayan et al., 2016).
6. Sound Mesial and distal neighboring teeth.
7. At least 6 natural teeth remaining in the same arch .
8. Mouth opening ≥ 30mm.
9. Thick phenotype.

Exclusion Criteria:

1. Poor oral hygiene condition.
2. Pregnant and lactating females.
3. Smokers.
4. Vulnerable groups (Prisoners and handicaps).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score | Baseline, 1,2 and 3 months after implantation.
  The Pink Esthetic Score is used to evaluate the soft tissue esthetics around single-tooth implants.
  It includes 7 parameters: mesial and distal papilla, tissue contours, gingival level, alveolar process, and both the color and texture of the soft tissue. Each is scored from 0 to 2, with higher scores reflecting more natural esthetics. For the papillae, a score of 0 indicates the papilla is missing, 1 is incomplete, and 2 is complete. Tissue contours are rated as unnatural (0), virtually natural (1), or natural (2). Gingival level is assessed based on vertical discrepancy with adjacent teeth: more than 2 mm scores 0, 1-2 mm scores 1, and less than 1 mm scores 2. The alveolar process is scored as clearly resorbed (0), slightly resorbed (1), or showing no difference (2). Finally, both soft tissue color and texture are evaluated against the neighboring tissue: a clear difference (0), a slight difference (1),no difference (2). The maximum PES is 14, represents ideal soft tissue esthetics.
Papilla index | baseline, 1,2 and 3 months
  The Papilla Index is a clinical tool used to evaluate the degree of interdental papilla fill in the proximal space around implants.
  It is scored on a scale from 0 to 4. A score of 0 indicates that no papilla is present. A score of 1 means less than half of the papilla height is visible. A score of 2 is assigned when half or more of the papilla height is present, though not completely filling the space.
  A score of 3 denotes a papilla that fully occupies the entire proximal space, representing the ideal scenario.
  A score of 4 indicates a hyperplastic papilla, where the tissue extends beyond the normal contours.

SECONDARY OUTCOMES:
Biochemical assessment of IL-1β level in the gingival crevicular fluid | After 2 months of implant placement
  Biochemical assessment of IL-1β level in the gingival crevicular fluid using Periopaper strip.

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel G Salem, Lecturer, Study Director — Faculty of Dentistry - Ain Shams University; Nevine H Kheir El Din, Professor, Study Director — Faculty of Dentistry - Ain Shams University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Abaseya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Pendleton N, Clague JE, Horan MA, Rabbitt PM, Jones M, Coward R, Lowe C, McInnes L. Concordance of Cornell medical index self-reports to structured clinical assessment for the identification of physical health status. Arch Gerontol Geriatr. 2004 May-Jun;38(3):261-9. doi: 10.1016/j.archger.2003.10.005. PMID 15066312
- [Background] Lashkarizadeh N, Foroudisefat M, Abyari S, Mohammadi M, Lashkarizadeh L. Is It Safe to Reuse Healing Abutments? An Experimental Study on IL-1beta and TNF-alpha Cytokine Levels in Peri-Implant Crevicular Fluid. J Prosthodont. 2022 Jun;31(5):399-404. doi: 10.1111/jopr.13474. Epub 2022 Feb 19. PMID 34962679
- [Background] Kunrath MF, Gupta S, Lorusso F, Scarano A, Noumbissi S. Oral Tissue Interactions and Cellular Response to Zirconia Implant-Prosthetic Components: A Critical Review. Materials (Basel). 2021 May 25;14(11):2825. doi: 10.3390/ma14112825. PMID 34070589
- [Background] Khatri M, Bansal M, Puri K, Mehrotra S, Kumar A, Rehan M. Evaluation of the correlation between interleukin 1beta levels in peri-implant crevicular fluid as an adjunctive diagnostic marker with clinical and radiographic parameters for assessing the peri-implant health status. Natl J Maxillofac Surg. 2022 Sep-Dec;13(3):421-429. doi: 10.4103/njms.njms_337_21. Epub 2022 Dec 10. PMID 36683945
- [Background] Chokaree P, Poovarodom P, Chaijareenont P, Yavirach A, Rungsiyakull P. Biomaterials and Clinical Applications of Customized Healing Abutment-A Narrative Review. J Funct Biomater. 2022 Dec 10;13(4):291. doi: 10.3390/jfb13040291. PMID 36547551
- [Background] Beretta M, Poli PP, Pieriboni S, Tansella S, Manfredini M, Cicciu M, Maiorana C. Peri-Implant Soft Tissue Conditioning by Means of Customized Healing Abutment: A Randomized Controlled Clinical Trial. Materials (Basel). 2019 Sep 19;12(18):3041. doi: 10.3390/ma12183041. PMID 31546800
- [Background] Bannunah AM. Biomedical Applications of Zirconia-Based Nanomaterials: Challenges and Future Perspectives. Molecules. 2023 Jul 15;28(14):5428. doi: 10.3390/molecules28145428. PMID 37513299
- [Background] Baltayan S, Pi-Anfruns J, Aghaloo T, Moy PK. The Predictive Value of Resonance Frequency Analysis Measurements in the Surgical Placement and Loading of Endosseous Implants. J Oral Maxillofac Surg. 2016 Jun;74(6):1145-52. doi: 10.1016/j.joms.2016.01.048. Epub 2016 Feb 1. PMID 26917203
- [Background] Almadani, T. M., Amer, A.-F. M., Abdallah, H. M., & El Sayed, I. S. Clinical and radiographic evaluation of peri-implant tissue changes associated with use of standard versus customized healing abutments. Al-Azhar Journal of Dental Science (2023), 26(2), 229-239.
- [Background] Ramenzoni LL, Fluckiger LB, Attin T, Schmidlin PR. Effect of Titanium and Zirconium Oxide Microparticles on Pro-Inflammatory Response in Human Macrophages under Induced Sterile Inflammation: An In Vitro Study. Materials (Basel). 2021 Jul 27;14(15):4166. doi: 10.3390/ma14154166. PMID 34361359

DOCUMENTS (1):
  • Study Protocol (2025-01-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT07095881/Prot_000.pdf